CLINICAL TRIAL: NCT05403177
Title: Marathon of Hope Cancer Centres Network Study for Ontario (MOHCCN-O)
Acronym: MOHCCN-O
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Ontario Institute for Cancer Research (Other); Terry Fox Research Institute (Other); Queen's University, Kingston, Ontario (Other); Ottawa Hospital Research Institute (Other); Queen's University (Other)
Responsible Party: Sponsor
Other Study IDs: MOHCCN-O
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Colorectal Cancer; Pancreas Cancer; Kidney Cancer; Prostate Cancer; Ovary Cancer; Head and Neck Cancer; Leukemia; Lymphoma; Lung Cancer; Melanoma; Solid Tumor
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Kidney Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms; Head and Neck Neoplasms; Leukemia; Lymphoma; Lung Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissues and blood samples will be collected from patients who are enrolled.
  Biopsy - up to 6 cores of tumour samples (1 time only) Blood - 20 mL collected in 2 x 10mL tubes (1 time only) Requesting archival: 10 x 10 um plus 1 H&E of Formalin-fixed paraffin embedded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MOHCCN-O: Tumor tissue and blood samples will be collected from patients who are enrolled in this study but do not yet have the molecular profiling data that are required to meet the gold standard criteria. Data will include: pathology, clinical biomarkers, imaging diagnostic information, whole genome and epi-genome sequencing of tumor and normal tissues, immunoprofiling of tumor tissues and/or peripheral blood, bioinformatic annotation of molecular information, and longitudinal clinical and outcome data.

SUMMARY:
The Marathon of Hope Cancer Centres Network (MOHCCN) is a national network of cancer centres that pursue collaborative cancer research in precision medicine (an emerging approach for disease treatment and prevention that considers individual variability in DNA, environment and lifestyle) to accelerate the discovery of innovations and improve the health outcomes for cancer patients

DETAILED DESCRIPTION:
The purpose of this study is to use evolving technologies such as genomics and artificial intelligence to study cancer so that the right treatment can be given to the right patient, at the right time. Approximately 15,000 participants will take part in the greater MOHCCN study across Canada in the first 5 years, and ultimately the goal is to enroll up to 100,000 over next 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological and/or cytological confirmation of blood or solid tumor malignancies. For tumour types where pre-surgical biopsy is not routinely performed to confirm a pathologic diagnosis of cancer, patients may consent to this protocol, but eligibility must be confirmed after pathology is finalized demonstrating presence of malignancy
2. All patients must be able to satisfy the required minimum data elements for the 15k gold standard cohort through:

   1. Already existing data that satisfies the minimal requirements of a gold standard case (refer to Table 1)
   2. Have sufficient biospecimens (tumor and/or blood samples) available for more comprehensive molecular and immunophenotypic characterization
3. Patients who do not satisfy the required minimum data elements but would like to participate, maybe requested to donate blood and undergo a fresh biopsy if the archived Formalin-fixed paraffin-embedded (FFPE) samples are not available, or in cases where a fresh tumor biopsy is deemed necessary for molecular profiling.
4. Participating patients must agree to share their anonymized clinical and genomic data

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any cancer patient
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients included in a pan-Canadian cohort with comprehensive clinical and genomic data | 5 years
  Consolidate and annotate data from patients included in a pan-Canadian cohort

SECONDARY OUTCOMES:
Development of standard practices to create a unique shareable dataset of molecular, imaging, clinical and health outcome information on Canadian cancer cases | 5 years
  Improve the cancer research paradigm by bringing teams or researchers together and leverage valuable information genomic and clinical data from Canadian cancer cases.
Clinical effectiveness and cost-effectiveness of precision cancer medicine to advance clinical implementation and reimbursement decisions | 5 years
  Health technology assessment tools will be used to evaluate the real-world value of precision medicine
Development and collection of patient-reported outcomes to enhance patient-centeredness in precision cancer medicine | 5 years
  Health technology assessment tools will be used to evaluate the real-world value of precision medicine

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario